CLINICAL TRIAL: NCT06963723
Title: Longitudinal Screening for Financial Hardship to Improve Outcomes in Patients With Advanced Cancer
Acronym: PROOF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alliance Foundation Trials, LLC. (Other)
Collaborators: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A232403
Record Dates: First submitted 2025-04-01; First posted 2025-05-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-03

CONDITIONS: Advanced Cancer; Metastatic Cancer
Keywords: Financial Toxicity
MeSH Terms: conditions — Neoplasm Metastasis; Financial Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants randomized to the intervention arm will complete their monthly screening using the single-item screening question (every 4 weeks for 12 months).
  Interventions: Other: Financial Hardship Screening
- Enhanced Usual Care (Active Comparator): Participants randomized to receive enhanced usual care will not be systematically screened for financial hardship through the electronic PRO Core system.
  Interventions: Other: Enhanced Usual Care

INTERVENTIONS:
Other: Financial Hardship Screening — Financial Hardship Screening and Financial Needs Assessment
  Arms: Intervention
Other: Enhanced Usual Care — Enhanced Usual Care
  Arms: Enhanced Usual Care

SUMMARY:
The study aims to determine whether monthly remote digital financial hardship screening among adults with advanced/metastatic cancer, undergoing outpatient systemic therapy with non-curative intent, improves patient-centered outcomes, including financial worry, health-related quality of life (HRQoL), symptom burden, patient-reported cancer treatment adherence, and exploratory outcomes of overall survival, patient-reported economic burden, patient-reported support received, patient-reported financial coping strategies, and health insurance literacy.

DETAILED DESCRIPTION:
Financial hardship is a common problem that affects patients treated for advanced cancer and leads to poor outcomes related to financial worry, health related quality of life (HRQoL), symptom burden, treatment adherence, and overall survival. Prior studies have shown that financial navigation may be an effective strategy to attenuate the impact of financial hardship. However, patients and clinicians have identified communication as a key barrier that prevents patients from being connected to sources of financial assistance. To address this critical gap in patient care, and based on strong preliminary data that financial hardship screening may improve patient outcomes, this financial hardship screening intervention will help connect patients to financial navigation resources. It is hypothesized that by connecting patients experiencing financial hardship with financial navigation resources, this intervention will lead to improved patient-centered outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Minimum age of 21
2. Understands English and/or Spanish
3. Has a diagnosis of advanced/metastatic cancer
4. Currently undergoing systemic therapy (enteral or parenteral) with non-curative intent
5. Has been receiving treatment for at least 2 months
6. Life expectancy of at least 6 months, in the opinion of the treating oncologist
7. Cognitively able to give informed consent

Exclusion Criteria:

1. Under the age of 21
2. Does not understand English or Spanish
3. Has cognitive deficits that would preclude understanding of consent form and/or questionnaires
4. Undergoing treatment with curative intent (e.g., adjuvant chemotherapy for breast, lung, or ovarian cancer, primary curative therapy for testis cancer or lymphoma)
5. Not undergoing systemic therapy (enteral or parenteral) with non-curative intent
6. Receiving treatment for fewer than 2 months
7. Life expectancy is less than 6 months, in the opinion of the treating oncologist

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2028-10-01 (Estimated); Study Completion 2029-04-01 (Estimated)

PRIMARY OUTCOMES:
Financial Worry | 6 months
  Patient-reported financial worry will be measured by the Functional Assessment of Chronic Illness Therapy-Comprehensive Score for Financial Toxicity (FACIT-COST) total scale.
  Possible score range: 0 to 44, with higher scores indicating better outcomes

SECONDARY OUTCOMES:
Health-related quality of life | 6 months
  Patient-reported health-related quality of life will be measured by the Functional Assessment of Cancer Therapy-General (FACT-G) total scale.
  Possible score range: 0 to 108, with higher scores indicating better outcomes
Symptom burden | 6 months
  Patient-reported symptom burden will be measured by the Functional Assessment of Cancer Therapy-General (FACT-G) physical well-being scale.
  Possible score range: 0 to 28, with higher scores indicating better outcomes
Cancer treatment adherence | 6 months
  Patient-reported cancer treatment adherence will be measured by the Domains of Subjective Extent of Nonadherence-Cancer (DOSE-Nonadherence-Cancer) extent of nonadherence scale, with patients classified as adherent (i.e., all responses of "none of the time" on the DOSE-Nonadherence-Cancer items for missing, skipping, or not taking a dose of medicine) versus nonadherent

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Blinder, MD, MSc, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - New Hampshire Oncology-Hematology, PA, Concord, New Hampshire
  - Solinsky Center for Cancer Care, Manchester, New Hampshire

IPD SHARING:
Plan to Share IPD: No